CLINICAL TRIAL: NCT06979505
Title: Dose-ranging Double-blind, Placebo-controlled Phase 2 Trial of GV101 for Weight Loss in Healthy Obese Participants
Brief Title: GV101 in Healthy Obese Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Graviton Bioscience Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GBS-201
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Weight Management

STUDY DESIGN:
Intervention Model Description: 1:1:1 random assignment to GV101 low dose, high dose, or matched placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GV101 low dose (Experimental)
  Interventions: Drug: GV101
- GV101 high dose (Experimental)
  Interventions: Drug: GV101
- GV101 matched placebo (Placebo Comparator)
  Interventions: Drug: GV101 placebo

INTERVENTIONS:
Drug: GV101 — GV101 suspension
  Arms: GV101 high dose; GV101 low dose
Drug: GV101 placebo — GV101 placebo suspension
  Arms: GV101 matched placebo

SUMMARY:
The purpose of this trial is to evaluate the efficacy and safety of GV101 for weight loss over a range of doses in participants with obesity. The primary efficacy endpoint is the mean percent change in body weight from baseline at Week 16 in each treated group as compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 18 years and ≤ 70 years with BMI ≥ 30.0 kg/m2 and ≤ 45.0 kg/m2 at the time of informed consent.
2. Willing and able to provide written informed consent to participate in the trial, available for all visits, and able and willing to comply with all trial procedures.
3. Except for obesity, otherwise healthy, as determined by the Investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, and ECGs at screening.
4. Have a stable body weight (< 3 kg self-reported change during the previous 90 days) before screening.
5. Willing to refrain from drastic changes in diet and physical activity regimen (those recommended via lifestyle counseling are acceptable).
6. Participants of reproductive potential (any male who has not undergone vasectomy more than 6 months prior to the first dose of investigational medicinal product [IMP] and any female who has not undergone bilateral oophorectomy, hysterectomy, total abdominal hysterectomy with bilateral salpingo-oophorectomy, bilateral tubal occlusion or ligation or who is not postmenopausal (a. A woman ≥55 years old not on hormone therapy, with amenorrhea for ≥12 months without an alternative medical cause, or b. A woman at least 55 years of age with a diagnosis of menopause prior to starting hormone replacement therapy or c. A woman > 40 and < 55 years of age with an intact uterus, not on hormone therapy, who has cessation of menses for at least r1 year without an alternative cause, AND a follicle-stimulating hormone (FSH) >25 mIU/mL or d. A woman with premature ovarian failure confirmed by historical FSH levels in the postmenopausal range prior to initiating HRT, or by a documented irreversible medical condition causing permanent infertility.)), who are heterosexually active, must agree to use a combination of two of the following methods of contraception (males must ensure their partner(s) use at least one method below to ensure at least two contraceptive methods are in place and must continue with this contraceptive plan for 90 days after the last dose of IMP; females must continue with this contraceptive plan for 28 days)
7. Male participants with a pregnant partner (including those who have undergone a vasectomy) must agree to use a condom from the first dose of the IMP administration until at least 90 days after the last (if applicable) dose of the IMP.
8. Male participants must agree not to donate sperm until 90 days after the last dose of IMP.

Exclusion Criteria:

1. Pregnant or lactating.
2. History of significant allergic reaction (e.g., immediate hypersensitivity, significant respiratory and skin symptoms such as Steven Johnson syndrome) or hypersensitivity to any drug.
3. History of clinically significant gastrointestinal disease or surgery that may affect IMP absorption. A history of appendectomy or cholecystectomy is not exclusionary.
4. Clinically significant physical examination abnormalities or clinically significant laboratory abnormalities at screening.
5. Obesity induced by other endocrinologic disorder (e.g., Cushing's syndrome).
6. Previous surgical treatment for obesity (excluding liposuction, if performed > 1 year before trial entry) and/or participants with recent (within 6 months) or planned endoscopic treatment for obesity.
7. Current or history (within 90 days before screening) of treatment with medications that may cause significant weight gain or loss, including systemic corticosteroids (except for a short course of treatment, i.e., 7 - 10 days), tricyclic antidepressants, atypical antipsychotics and mood stabilizers (e.g., imipramine, amitriptyline, mirtazapine, paroxetine, phenelzine, chlorpromazine, thioridazine, clozapine, olanzapine, valproic acid and its derivatives, and lithium).
8. Current participation (or within the last 90 days) in an organized weight reduction program or currently using or used within 90 days before screening: pramlintide, sibutramine, orlistat, zonisamide, topiramate, phentermine, naltrexone, bupropion, lorcaserin, metformin, or any GLP-1R and/or glucose-dependent insulinotropic polypeptide (GIP) agonists (either by prescription or as part of a clinical trial).
9. Evidence of clinically significant hepatic or renal impairment, including but not limited to screening test results of ALT and AST above 1.5x the ULN, total bilirubin above the ULN, history of Gilbert's syndrome or of elevated bilirubin, especially while fasting.
10. History of clinically significant QTcF interval prolongation, or a QTcF interval of > 470 ms in females or of > 450 ms in males at screening.
11. Clinically significant vital sign abnormalities at screening (systolic blood pressure [SBP] < 90 or > 150 mm Hg, diastolic blood pressure [DBP] < 50 or > 100 mm Hg, or heart rate [HR] < 50 or > 100 bpm). Retesting is allowed at the discretion of the site Investigator or designee.
12. Not willing to limit alcohol consumption to 2 drinks per day for males and 1 drink per day for females. History of alcohol misuse within 1 year prior to screening or regular alcohol consumption (more than 14 units per week [1 unit = 150 mL wine, 360 mL beer, or 45 mL 40% alcohol]) within 6 months prior to the screening visit.
13. History of illicit drug misuse within 1 year prior to screening, or use of hard drugs (e.g., cocaine, phenylcyclohexyl piperidine [PCP], crack, opioid derivatives, and amphetamine derivatives) within 1 year prior to screening. A history of marijuana or tetrahydrocannabinol (THC)- product use within 30 days of enrollment and unwillingness to abstain from marijuana or the use of THC-containing products during the trial is also exclusionary. Stable daily CBD use is allowed (stable for > 30 days prior to randomization and planned continued stable use throughout the trial). Intermittent CBD use is not allowed.
14. Participation in a clinical trial involving the administration of an investigational or marketed drug or device use within 30 days or 5 half-lives, whichever is longer, before IMP administration; administration of a biological product in the context of a clinical trial within 90 days or 5 half-lives before IMP administration, whichever is longer, or concurrent participation in an experimental trial that does not involve the administration of an IMP or device use.
15. Not willing to refrain from strenuous exercise or vigorous activity (e.g., heavy lifting, weight training, yard work in hot weather, and aerobics) for 72 hours before each blood collection for clinical laboratory tests.
16. Use of drugs and foods including CYP3A4 inhibitors or inducers (Table 10), UGT1A1 substrates and inhibitors, daily use of medications that are substrates of CYP2C8, CYP2C9, or CYP2C19 and have a narrow therapeutic index.
17. The following test results:

    1. Positive hepatitis B, positive hepatitis C Ab with non-negative HCV RNA test, or positive HIV test at screening
    2. Calculated estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 at screening
    3. Positive pregnancy test at any time from screening onwards
    4. Positive drug test at screening
    5. HbA1c ≥ 6.5% and/or known history of type 1 or type 2 diabetes mellitus, other forms of diabetes like LADA, MODY and secondary diabetes.

       Note: Patients with h/o gestational diabetes (but no diagnosis of T2DM post partum) can qualify.
    6. Thyroid stimulating hormone (TSH) > 6 mIU/L or < 0.4 mIU/L at screening
    7. Fasting triglycerides ≥ 5.65 mmol/L (i.e., 500 mg/dL)
    8. ALT or AST above 1.5x the ULN, total bilirubin above the ULN at screening
    9. Platelet count < 150,000 platelets/mL
18. Participant unwilling or unable to abstain from using nicotine or tobacco, cigars, cigarettes, e-cigarettes/vaping, pipes, or nicotine patches for 45 minutes prior to trial visits.
19. History or evidence of any other clinically significant disorder, condition, or disease or any other reason that, in the opinion of the Investigator or physician, would pose a risk to participant safety or interfere with the trial evaluation, procedures, or completion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-01-28 (Actual); Study Completion 2026-01-28 (Actual)

PRIMARY OUTCOMES:
Mean percent change in body weight from baseline at Week 16 in each treated group as compared with placebo | 16 weeks

CONTACTS AND LOCATIONS:
Locations (20):
- United States (16):
  - Lakeview Clinical Research, LLC, Guntersville, Alabama
  - Arizona Clinical Trials, Tucson, Arizona
  - Catalina Research Institute, LLC, Montclair, California
  - Encompass Clinical Research, Spring Valley, California
  - Louisville Metabolic and Atherosclerosis Research Center (L-MARC), Louisville, Kentucky
  - Tandem Clinical Research, Marrero, Louisiana
  - Study Metrix Research, City of Saint Peters, Missouri
  - Kansas City Research Institute, Kansas City, Missouri
  - Mercury Street Medical, Butte, Montana
  - Hassman Research Institute, Berlin, New Jersey
  - Coastal Research Institute, LLC, Fayetteville, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - Velocity Clinical Research - Cleveland, Cleveland, Ohio
  - Velocity Clinical Research - Dallas, Dallas, Texas
  - Advanced Research Institute - Ogden, Ogden, Utah
  - Chrysalis Clinical Research, St. George, Utah
- Israel (4):
  - Hadassah Medical Center Ein Karem, Jerusalem, Israel
  - Hasharon Hospital, Petah Tikva, Israel
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva, Israel
  - Sheba Medical Center, Tel Litwinsky, Israel